CLINICAL TRIAL: NCT01151748
Title: Intra-arterial Chemotherapy for Advanced Intraocular Retinoblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study abandoned; Could not obtain final SRC approval due to IND disagreements
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDSEYE0001; SU-07072009-3000 (Other: Stanford University)
Record Dates: First submitted 2010-03-04; First posted 2010-06-28 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Retinoblastoma; Eye Cancer
MeSH Terms: conditions — Retinoblastoma; Eye Neoplasms

INTERVENTIONS:
Procedure: Intra-arterial infusion of chemotherapy

SUMMARY:
Phase II study of selective intra-arterial infusion of chemotherapy for intraocular retinoblastoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with advanced intraocular retinoblastoma (International Retinoblastoma Classification group D or E*).
2. Patients with tumor recurrence or vitreous seeding following completion of systemic chemotherapy or previous radiation therapy.

Exclusion Criteria:

1. Congenital brain anomaly identified on MRI.
2. History of systemic coagulopathy.
3. Evidence of extra ocular retinoblastoma on clinical examination or neuroimaging.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Response: Globe salvage rate (Eyes saved/Eyes treated). This will be determined by clinical ocular examination. | Follow-up will be performed for one year from treatment date.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Kim, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States